CLINICAL TRIAL: NCT00040885
Title: Docetaxel And Infliximab/Placebo In Non-Small Cell Lung Cancer (NSCLC) Patients Greater Than Or Equal To 65 Years Of Age Or In NSCLC Patients With Poor Performance Status: A Double-Blind Randomized, Placebo-Controlled Trial To Prevent And Treat Wasting, Anorexia, And Asthenia In Chemotherapy-Naive And Previously-Treated Patients
Brief Title: Docetaxel With or Without Infliximab in Treating Weight Loss, Loss of Appetite, and Fatigue in Patients With Unresectable Non-Small Cell Lung Cancer (Infliximab Treatment Discontinued Effective 10/05/05)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N01C9; NCI-2012-02472 (Registry Identifier: CTRP (Clinical Trials Reporting System)); NCI-P02-0226; CDR0000069417 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Anorexia; Cachexia; Fatigue; Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; fatigue; anorexia; cachexia
MeSH Terms: conditions — Anorexia; Cachexia; Fatigue; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Infliximab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- infliximab + docetaxel (Experimental): Patients receive infliximab IV over 2 hours once weekly on weeks 1, 3, and 5 of the first course and once weekly on weeks 1 and 5 of all subsequent courses and docetaxel IV over 1 hour (immediately after completion of infliximab infusion once weekly on weeks 1-6 of each course.
  Treatment repeats every 8 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity.
  Quality of life, fatigue, appetite/anorexia, cachexia, and weight are assessed at baseline, weekly on weeks 1-8, and then monthly for the remainder of study treatment.
  Patients are followed every 6 months for 5 years.
  Interventions: Biological: infliximab; Drug: docetaxel
- placebo + docetaxel (Active Comparator): Patients receive docetaxel IV over 1 hour (immediately after completion of infliximab infusion once weekly on weeks 1-6 of each course. Patients receive placebo IV over 2 hours once weekly on weeks 1, 3, and 5 of the first course and once weekly on weeks 1 and 5 of all subsequent courses.
  Treatment repeats every 8 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity.
  Quality of life, fatigue, appetite/anorexia, cachexia, and weight are assessed at baseline, weekly on weeks 1-8, and then monthly for the remainder of study treatment.
  Patients are followed every 6 months for 5 years.
  Interventions: Drug: docetaxel; Other: placebo

INTERVENTIONS:
Biological: infliximab
  Arms: infliximab + docetaxel
Drug: docetaxel
Other: placebo
  Arms: placebo + docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Infliximab may improve cancer-related weight loss, lack of appetite, and fatigue. It is not yet known whether docetaxel is more effective with or without infliximab in preventing weight loss and fatigue in patients with advanced cancer. (Infliximab treatment discontinued effective 10/05/05)

PURPOSE: Randomized phase III trial to determine the effectiveness of docetaxel with or without infliximab in preventing weight loss, loss of appetite, and fatigue in patients who have unresectable non-small cell lung cancer. (Infliximab treatment discontinued effective 10/05/05)

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the improvement or stabilization of weight in elderly or poor performance status patients with unresectable non-small cell lung cancer treated with docetaxel with or without infliximab (infliximab treatment discontinued effective 10/05/05).
* Compare appetite and functional status in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the augmentation or maintenance of lean tissue in patients treated with these regimens.
* Compare the response rates and time to disease progression in patients treated with these regimens.
* Compare the survival of patients treated with these regimens.
* Determine whether the tumor necrosis factor-alpha polymorphisms in the -308 and -238 regions predict which cancer patients will experience loss of appetite and weight and which patients might potentially benefit from infliximab (infliximab treatment discontinued effective 10/05/05).

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to weight loss within the past 6 months (0% vs more than 0% to less than 5% vs at least 5%), number of prior chemotherapy regimens (0 vs 1 vs more than 1), gender, and GBU prognostic index (good vs bad vs unsure).

* Part A (non-randomized, single-center portion of study): Five patients receive infliximab IV (infliximab treatment discontinued effective 10/05/05) over 2 hours once weekly on weeks 1, 3, and 5 of the first course and once weekly on weeks 1 and 5 of all subsequent courses and docetaxel IV over 1 hour (immediately after completion of infliximab infusion [infliximab treatment discontinued effective 10/05/05]) once weekly on weeks 1-6 of each course. Treatment repeats every 8 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity.

If none of the 5 patients experiences any grade 4 or 5 toxicity directly attributable to infliximab (infliximab treatment discontinued effective 10/05/05), additional patients are accrued for part B of the study.

* Part B (randomized, multicenter portion of study): Patients are randomized to 1 of 2 treatment arms.

  * Arm I (infliximab treatment discontinued effective 10/05/05): Patients receive infliximab and docetaxel as in part A.
  * Arm II: Patients receive docetaxel as in part A and placebo IV over 2 hours according to the infliximab schedule in part A (infliximab treatment discontinued effective 10/05/05).

Treatment in both arms repeats as in part A.

Quality of life, fatigue, appetite/anorexia, cachexia, and weight are assessed at baseline, weekly on weeks 1-8, and then monthly for the remainder of study treatment.

Patients are followed every 6 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable non-small cell lung cancer that is considered incurable with other therapies
* Chemotherapy naive or previously treated disease
* Meets one of the following criteria:

  * Age 65 and over with ECOG performance status of 0-2
  * Under age 65 with ECOG performance status of 2
* No symptomatic or known untreated brain metastases

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics
* Adult

Performance status:

* See Disease Characteristics
* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST and/or ALT ≤ 2.5 times upper limit of normal (ULN) if alkaline phosphatase less than ULN OR
* Alkaline phosphatase ≤ 4 times ULN if ALT less than ULN
* No ascites

Renal:

* Creatinine ≤ 1.5 times ULN

Cardiovascular:

* No prior or concurrent congestive heart failure

Pulmonary:

* No prior tuberculosis or positive purified protein derivative skin test (tuberculin test)

Other:

* No prior anaphylactic reaction to any taxane
* No known mechanical obstruction of the alimentary tract, malabsorption, or intractable vomiting (more than 5 episodes per week)
* No infection or chronic debilitating illness that would increase the risk of chemotherapy administration
* No grade 2 or greater peripheral neuropathy of any etiology
* No edema
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer
* Alert and mentally competent
* Able to complete questionnaires alone or with assistance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior docetaxel for metastatic non-small cell lung cancer

Endocrine therapy:

* At least 1 month since prior adrenal steroids, androgens, progestational agents, or appetite stimulants
* No concurrent adrenal steroids, androgens, progestational agents, or appetite stimulants unless needed (e.g., steroids for CNS metastases)
* Concurrent inhaled, topical, or optical steroids allowed
* Concurrent short-term dexamethasone around days of chemotherapy administration allowed for protection against anaphylaxis and emesis

Radiotherapy:

* More than 3 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow

Surgery:

* More than 3 weeks since prior major surgery

Other:

* More than 3 weeks since other prior antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2002-10; Primary Completion 2006-02 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Assessment of weight | Up to 5 years
Rate of weight change | Up to 5 years

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
Incidence of treatment-related toxicity | Up to 5 years
Cancer-related fatigue as measured by the Brief Fatigue Inventory | Up to 5 years
Time-to-weight decline | Up to 5 years
Appetite | Up to 5 years
Lean tissue changes | Up to 5 years
Quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (188):
- United States (188):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thorton, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Alegent Health Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Health Center, Onawa, Iowa
  - Ottumwa Regional Health Center Cancer Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Adult and Pediatric Urology, P.L.L.P., Saint Cloud, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Fremont Area Medical Center, Fremont, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - United States Air Force Medical Center Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Luther Mildelfort Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Result] Jatoi A, Ritter HL, Dueck A, Nguyen PL, Nikcevich DA, Luyun RF, Mattar BI, Loprinzi CL. A placebo-controlled, double-blind trial of infliximab for cancer-associated weight loss in elderly and/or poor performance non-small cell lung cancer patients (N01C9). Lung Cancer. 2010 May;68(2):234-9. doi: 10.1016/j.lungcan.2009.06.020. Epub 2009 Aug 8. PMID 19665818